CLINICAL TRIAL: NCT03095885
Title: A Pilot Study of Oxalate Absorption in Secondary Hyperoxaluria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALLN-177-204
Record Dates: First submitted 2017-03-20; First posted 2017-03-30 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Secondary Hyperoxaluria; Nephrolithiasis; Hyperoxaluria; Kidney Stones
Keywords: Urine Oxalate; Nephrolithiasis; Kidney Stones; Hyperoxaluria; Enteric Hyperoxaluria; urological Diseases; Kidney Diseases; Dietary Oxalate; Idiopathic Hyperoxaluria; Oxalate Absorption
MeSH Terms: conditions — Nephrolithiasis; Hyperoxaluria; Kidney Calculi; Urologic Diseases; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test Meal (Other): controlled oxalate-rich test meal
  Interventions: Other: Test Meal

INTERVENTIONS:
Other: Test Meal

SUMMARY:
Identify individuals with greater absorption of oxalate based on increase in urinary oxalate excretion in response to a controlled oxalate-rich test meal.

DETAILED DESCRIPTION:
This was a prospective 4-day study of oxalate absorption in subjects with secondary hyperoxaluria. Subjects visited the research center three times for outpatient visits (Screening, Test Day 3, Day 4).

Subjects were instructed to follow a low-oxalate diet, consuming only study-specified food choices that had low or no oxalate and controlled calcium content Days 1 through 4 (Baseline Period through the Day 4 clinic visit) and, on Test Day 3, consumed an oxalate-rich test meal.

Subjects performed three 24-hour urine collections during Screening, Baseline Day 2, and Test Day 3. Test Day 3 included the oxalate-rich test meal and the subject collected a 24-hour urine separated into 4 urine collection intervals. (Pre-test meal, post-test meal to 4 hours, 4-6 hours post test meal and remaining time to complete 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant and non-lactating females
* History of hyperoxaluria secondary to a known underlying enteric disease (e.g., Crohn's disease, bariatric surgery, and others) or without a known underlying cause (idiopathic), and kidney stones.
* Urinary oxalate ≥ 40 mg of oxalate/24 hr at screening.
* If taking drugs for the prevention of stone disease, including pyridoxine, thiazides (chlorthalidone, hydrochlorothiazide, and indapamide), citrate supplements, and allopurinol, there must have been no changes in these medications for at least one month prior to screening and no changes are anticipated for the duration of the study.
* Able to understand and provide written informed consent.

Exclusion Criteria:

* Under or over-collection on screening 24-hour urine collection (mg creatinine/kg body weight outside of gender-specific range).
* Estimated glomerular filtration rate (eGFR) <40 mL/minute/1.73 m^2 or acute renal failure.
* Primary hyperoxaluria.
* Allergy, intolerance, or any other factors limiting ability to consume the study foods or adhere to the study meal schedule.
* Positive pregnancy test during Screening.
* Clinically significant findings (including acute renal colic), an ongoing clinically significant illness requiring changes in management, or any planned medical/surgical procedure during the study.
* Malignancy undergoing active therapy; patients in remission on chronic suppressive or maintenance therapies are not excluded.
* Investigational compound within 30 days prior to screening.
* Investigator determined that the subject would not be able to adhere or to complete the study procedures , or could not discontinue Vitamin C supplements, calcium supplements, or other medications that could interfere with oxalate absorption and/or excretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Kausz, MD, MS, Study Director — Allena Pharmaceuticals
Locations (5):
- United States (5):
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Applied Research Center of Arkansas, Inc., Little Rock, Arkansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - Omega Medical Research, Warwick, Rhode Island
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Meal
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Set: The Enrolled Set included all subjects who were determined to be eligible for the study after screening assessments and were enrolled in the study.
Arm/Group | Enrolled Set
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.45 (8.04)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/minute/1.73 /m^2] | 80.7 (17.4)
Hyperoxaluria Classification [Count of Participants; unit: Participants]
  Idiopathic Hyperoxaluria | 17
  Enteric Hyperoxaluria | 5
Number of Kidney Stone Episodes at Study Entry [Mean (Standard Deviation); unit: Episodes] | 5 (5.37)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Oxalate Absorption Normalized by Baseline Urinary Oxalate Excretion Over a 24 Hour Test Period
Description: Percent of oxalate absorption normalized by baseline was calculated by 100*[UOx/test - UOx/baseline]/Ox intake from the test meal.
Time Frame: 24 hours during baseline and test day following oxalate-rich meal
Population: Enrolled set which included all enrolled subjects
Measure: Mean (Standard Deviation); unit: percentage of oxalate absorption
Arm/Group | Test Meal
Number analyzed (Participants) | 22
percentage of oxalate absorption | 2.84 (2.36)

2. Secondary Outcome: Percent of Oxalate Absorption By Test Interval
Description: Percent of Oxalate absorption by test interval was calculated as the urinary oxalate excretions (mg) during the test interval divided by the amount of oxalate in the test meal.
Time Frame: 0-4 hours post test meal, 0-6 hours post test meal, 0-24 hours post test meal
Population: Enrolled set which included all enrolled subjects
Measure: Mean (Standard Deviation); unit: percentage of oxalate absorption
Arm/Group | Test Meal
Number analyzed (Participants) | 22
percentage of oxalate absorption
  0-4 Hours post test meal | 2.11 (0.52)
  0-6 hours post test meal | 3.55 (0.88)
  0-24 hours post test meal | 10.83 (3.04)

3. Secondary Outcome: Percent Change From Baseline for Urinary Oxalate to Creatinine Ratio by Test Interval
Description: Urinary oxalate (UOx) excretion was normalized to units of mg/g creatinine by dividing the UOx in mg by the creatinine value in g from the same collection. Percent change from baseline for UOx/Cr from Baseline was calculated by 100 * [UOx/Cr for the test interval - UOx/Cr at Baseline] / UOx/Cr at Baseline.
Time Frame: 24 hours during baseline, 0 to 4 hours post test meal, 0-6 hours post test meal, 6-24 hours post test meal, 0-24 hours post test meal
Population: Enrolled set which included all enrolled subjects
Measure: Mean (Standard Deviation); unit: Percentage of change of UOx/Cr
Arm/Group | Test Meal
Number analyzed (Participants) | 22
Percentage of change of UOx/Cr
  0-4 hours post test meal | 68.17 (93.05)
  0-6 hours post test meal | 84.73 (100.05)
  6-24 hours post test meal | 45.39 (62)
  0-24 hours post test meal | 47.14 (64.82)

ADVERSE EVENTS:
Time Frame: 34 days (adverse events were recorded from the time of informed consent until the last study visit, and the screening period was approximately 30 days)
Description: Since no investigational product was administered; no drug-related adverse events (AEs) occurred. The investigator assessed AEs by intensity (severity) and causality in relation to the study intervention, which was the study diet. Any untoward symptoms or worsening of medical conditions reported during the study were recorded as AEs.
Arm/Group | Test Meal
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Meal (N=22)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other